CLINICAL TRIAL: NCT00927940
Title: The Clinical Evaluation of the MDT-4107 Drug-Eluting Coronary Stent in De Novo Lesions in Native Coronary Arteries
Brief Title: RESOLUTE Japan - The Clinical Evaluation of the MDT-4107 Drug-Eluting Coronary Stent
Acronym: RJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Collaborators: Medtronic Japan Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT2-07-03
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Arterial Occlusive Diseases; Myocardial Ischemia; Cardiovascular Diseases; Coronary Artery Disease
Keywords: TARGET VESSEL REVASCULARIZATION (TVR); MYOCARDIAL INFARCTION (MI); TARGET VESSEL FAILURE (TVF); TARGET LESION REVASCULARIZATION (TLR); TARGET LESION FAILURE (TLF); STENT THROMBOSIS; RESTENOTIC LESION; PERCUTANEOUS CORONARY INTERVENTION (PCI)
MeSH Terms: conditions — Arterial Occlusive Diseases; Myocardial Ischemia; Cardiovascular Diseases; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug Eluting Stent (Experimental): All patients may have one or two lesions, if the two lesions are located in separate coronary arteries. A patient with one or two lesions treated with stents of diameter 2.5mm - 3.5mm will be designated in this study.
  Interventions: Device: MDT-4107 Drug Eluting Stent

INTERVENTIONS:
Device: MDT-4107 Drug Eluting Stent — Implantation of a MDT-4107 Zotarolimus-Eluting Coronary Stent
  Other Names: Zotarolimus Eluting Coronary Stent

SUMMARY:
The objective of the study is to verify the safety and efficacy of the MDT-4107 Drug-Eluting Coronary Stent for the treatment of de novo lesions in native coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable candidate for percutaneous coronary intervention (PCI),stenting, and emergency coronary artery bypass graft surgery
* Clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia and/or positive functional study
* Informed consent
* Patient agrees to comply with specified follow-up evaluations at same investigational site
* Single target lesion or two target lesions located in separate coronary arteries
* De novo lesion(s) in native coronary artery(ies)
* Target lesion(s) ≤ 27 mm in length
* Target vessel(s) have reference vessel diameter 2.5 mm to 3.5 mm

Exclusion Criteria:

* Within 7 days of implant platelet count <100,000 cells/mm³ or >700,000 cells/mm³; white blood cell (WBC) count <3,000 cells/mm³; serum creatinine level >2.5 mg/dl
* Acute myocadial infarction (MI) within 72 hrs of the index procedure (Q wave myocardial infarction(QWMI) or any elevation of Creatinine Kinase Mycocardial-band Isoemzyme (CK-MB) > lab upper limit of normal)
* Previous PCI of target vessel(s) within 9 months prior to the procedure
* Planned PCI of any vessel within 30 days post-index procedure and/or planned PCI of target vessel(s) within 12 months post-index procedure
* History of stroke or transient ischemic attack (TIA) within prior 6 months
* Participating in investigational drug/device study that has not completed primary endpoint or interferes with study endpoints
* Inability to comply with required trial antiplatelet regimen
* Previous stent in target vessel unless it has been at least 9 months since stent placed and target lesion(s) is/are at least 15 mm from previous stent
* Target vessel(s) has/have other lesions w/ > 40% diameter stenosis
* Unprotected left main coronary artery disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital
Locations (14):
- Japan (14):
  - Toyohashi Heart Center, Aichi
  - Hospital Hakodate Hokkaido, Hokkaido
  - Kansai Rosai Hospital, Hyōgo
  - Kanto Rosai Hospital, Kanagawa
  - Yokohama Tobu Hospital, Kanagawa
  - Shonan Kamakura General Hospital, Kanagawa
  - Kumamoto Rosai Hospital, Kumamoto
  - Kyoto Katsura Hospital, Kyoto
  - Kurashiki Central Hospital, Okayama
  - Jichi Medical University Hospital, Tochigi
  - The Cardiovascular Institute Hospital, Tokyo
  - Showa University Hospita, Tokyo
  - Toho University Medical Center, Ohashi Hospital, Tokyo
  - Teikyo University Hospital, Tokyo

REFERENCES:
- [Derived] Saito S, Maehara A, Vlachojannis GJ, Parise H, Mehran R; RESOLUTE Japan Investigators. Clinical and angiographic evaluation of the resolute zotarolimus-eluting coronary stent in Japanese patients - long-term outcome in the RESOLUTE Japan and RESOLUTE Japan small vessel study. Circ J. 2015;79(1):96-103. doi: 10.1253/circj.CJ-14-0836. Epub 2014 Nov 27. PMID 25428602
- [Derived] Silber S, Kirtane AJ, Belardi JA, Liu M, Brar S, Rothman M, Windecker S. Lack of association between dual antiplatelet therapy use and stent thrombosis between 1 and 12 months following resolute zotarolimus-eluting stent implantation. Eur Heart J. 2014 Aug 1;35(29):1949-56. doi: 10.1093/eurheartj/ehu026. Epub 2014 Feb 7. PMID 24510638
- [Derived] Silber S, Serruys PW, Leon MB, Meredith IT, Windecker S, Neumann FJ, Belardi J, Widimsky P, Massaro J, Novack V, Yeung AC, Saito S, Mauri L. Clinical outcome of patients with and without diabetes mellitus after percutaneous coronary intervention with the resolute zotarolimus-eluting stent: 2-year results from the prospectively pooled analysis of the international global RESOLUTE program. JACC Cardiovasc Interv. 2013 Apr;6(4):357-68. doi: 10.1016/j.jcin.2012.11.006. Epub 2013 Mar 20. PMID 23523454
- [Derived] Farooq V, Vranckx P, Mauri L, Cutlip DE, Belardi J, Silber S, Widimsky P, Leon M, Windecker S, Meredith I, Negoita M, van Leeuwen F, Neumann FJ, Yeung AC, Garcia-Garcia HM, Serruys PW. Impact of overlapping newer generation drug-eluting stents on clinical and angiographic outcomes: pooled analysis of five trials from the international Global RESOLUTE Program. Heart. 2013 May;99(9):626-33. doi: 10.1136/heartjnl-2012-303368. Epub 2013 Mar 6. PMID 23468513
- See also: Medtronic Clinical Trials Link — http://clinicaltrials.medtronic.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient and the last patient were enrolled on Mar. 23, 2009 and Oct. 30, 2009 respectively. Total 100 patients were enrolled in this study from 14 sites.
Groups:
- Zotalolimus Eluting Sttent: All patients may have one or two lesions, if the two lesions are located in separate coronary arteries. A patient with one or two lesions treated with stents of diameter 2.5mm - 3.5mm will be designated in this study.
Period: Overall Study
Arm/Group | Zotalolimus Eluting Sttent
Started | 100
Completed | 99 (A patient died before 30 days follow up. This pasitent is excluded from primary analysis.)
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zotalolimus Eluting Sttent
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 77
Region of Enrollment [Number; unit: participants]
  Japan | 100

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Lumen Loss (LLL)
Description: The difference between the post-procedure immediate minimal lumen diameter (MLD) and follow up angigraphy MLD
Time Frame: Post procedure, 8 Months
Population: Actually a patient was excluded from this analysis because of death before 30 days follow up.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Zotarolimus Eluting Stent: 100 lesion of 100 ITT patients were subjected for this analysis.
Arm/Group | Zotarolimus Eluting Stent
Number analyzed (Participants) | 99
mm | 0.13 (0.22)

2. Secondary Outcome: Percent of Patient With Target Lesion Failure(Major Secondary Endpoint)
Description: Major Secondary Endpoint Target lesion fature (TLF) is defined as cardiac death, target vessel myocardial infarction(Q wave and non-Q wave), or clinically-driven target lesion revascularization (TLR) by percutaneous or surgical methods.
Time Frame: 12 months
Population: ITT population
Measure: Number; unit: percentage of participants with TLF
Arm/Group | Zotarolims Eluting Stent
Number analyzed (Participants) | 100
percentage of participants with TLF | 4.0 [1.1 to 9.9]

3. Secondary Outcome: Success(Device, Lesion, Procedure), Major Adverse Cardiac Events (MACE), Target Vessel Failure (TVF), and Stent Thrombosis
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Rates of Incomplete Stent Apposition, Neointimal Hyperplastic Volume and Percent Volume Obstruction (%VO)
Time Frame: 8 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Zotalolimus Eluting Sttent
Serious Adverse Events (participants affected / at risk) | 35/100
Other Adverse Events (participants affected / at risk) | 58/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zotalolimus Eluting Sttent (N=100)
CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 5
CORONARY ARTERY STENOSIS (Cardiac disorders) | 3
ANGINA PECTORIS (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 1
MIOCARDIAL INFARCTION (Cardiac disorders) | 4
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
COLONIC POLYP (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 2
LOWER GASTROINTESTINAL HEAMORRAGE (Gastrointestinal disorders) | 2
MELAENA (Gastrointestinal disorders) | 1
PYREXIA (General disorders) | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1
DIVERTICULITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 2
C-REACTIVE PROTEIN INCREASED (Investigations) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RECTOSIGMOID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 1
DECREASED ACTIVITY (Psychiatric disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PERCUTANEOUS CORONARY INTERVENTION (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zotalolimus Eluting Sttent (N=100)
CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 6
STOMATISIS (Gastrointestinal disorders) | 5
CHEST DISCONFORT (General disorders) | 12
NASOPHARYNGITIS (Infections and infestations) | 12
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5
ASPARATATE AMINOTRANSFERASE INCREASED (Investigations) | 8
BLOOD CREATINE PHOPHOKINASE INCREASED (Investigations) | 15
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 6
BLOOD PRESSURE DECREASED (Investigations) | 5
BLOOD UREA INCREASED (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No